CLINICAL TRIAL: NCT01055561
Title: An Open-label Multi-center Safety and Tolerability Study of Acupuncture for Patients With Behavioural and Psychological Symptoms of Dementia & Healthy Volunteers
Brief Title: A Study of Acupuncture for Patients With Behavioural and Psychological Symptoms of Dementia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008SZ0135
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Acupuncture; Behavioral and Psychological Symptoms of Dementia; BPSD; MMSE; BEHAVE-AD; The Questionnaire of Acupuncture Events; healthy volunteers
MeSH Terms: conditions — Alzheimer Disease; Dementia; Behavior | interventions — Acupuncture Therapy; Complementary Therapies; Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients (Experimental)
  Interventions: Other: Acupuncture
- Healthy volunteers (Experimental)
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Participators will be stimulated at specific acupuncture points as determined for the disease by the professional acupuncturists, and acupuncture once a day,last for one week.
  Other Names: Complementary and Alternative Medicine; Traditional Chinese Medicine

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of acupuncture for patients with BPSD & healthy volunteers.

DETAILED DESCRIPTION:
This open label study is designed to evaluate the safety and tolerability of acupuncture as a intervention for patients with Behavioral and Psychological Symptoms of Dementia (BPSD)& healthy volunteers,and this study will enroll a total of 30(15 patients,15healthy volunteers) patients who are suffered from BPSD or healthy volunteers.The patients who have to be suitable for the standard of inclusion criteria will be included,and who have one condition of the exclusion criteria will be excluded,and so do the healthy volunteers.For each enrolled participant will obtain a baseline psychiatric and medical assessment, results of the Mini-Mental Status-Evaluation (MMSE),Behavioral Pathology in Alzheimer's Disease Rating Scale(BEHAVE-AD),Activity of Daily Living Scale(ADL)and other basic information prior to beginning acupuncture.For each participant will get acupuncture which once a day for 7 days running. During the trial the Questionnaire of Acupuncture-related Events have to be evaluated every day, and at the end of the intervention,all of the MMSE,BEHAV-AD,ADL and Treatment Emergent Symptom Scale (TESS)will be investigated.

ELIGIBILITY:
The eligibility criteria of the patients arm:

Inclusion Criteria:

1. patients who aged 60 to 85(inclusive) years
2. The MMSE score of patients must be between 5 to 26
3. Patients with diagnosis of Alzheimer's Disease according to DSM-Ⅳ（Diagnostic and Statistical Manual of Mental Disorders Fourth Edition)
4. patients have one or more "target symptoms" of Behavioral and Psychological Symptoms of Dementia(BPSD) on the behavioral psychology in Alzheimer's disease rating scale (BEHAVE-AD),and the "target symptoms " of BEHAVE-AD have to have occurred nearly daily during the previous week or at least intermittently for 4 weeks
5. Patients (or a legally acceptable representative)have signed the informed consent form

Exclusion Criteria:

1. Received a diagnosis of a primary psychotic disorder (e.g.schizophrenia，bipolar disorder, severe or recurrent depression),other dementia such as vascular dementia,complex dementia or Lewy-body dementia,or psychosis,agitation, or aggression that could be better accounted for by another medical condition, or substance abuse
2. Had severe system disease (e.g., cardiovascular, hepatorenal, hematopoietic system) or infectious disease
3. Received medication (e.g.,benzodiazepines, antipsychotics, or anticholinergics)which could treat BPSD within 2 weeks prior to the first acupuncture of the study
4. Participated in any clinical trial of drug within 4 weeks prior to the study
5. History of taking acupuncture

The eligibility criteria of the healthy volunteers arm:

Inclusion Criteria:

1. Healthy volunteers aged 60 to 85(inclusive) years who have provided written informed consent
2. MMSE> or =27
3. Have relative better health condition who do not suffered from severe system disease (e.g.,cardiovascular, hepatorenal, hematopoietic system) or infectious disease

Exclusion Criteria:

1. History of significant neurological (including history of seizures,EEG abnormalities or dementia) or psychotic disorder (e.g.schizophrenia，bipolar disorder, severe or recurrent depression)
2. History of drug or alcohol abuse
3. History of taking medication that may be impair the function of cognition or psychotic behavior within 4 weeks before the study
4. Participated in any clinical trial of drug within 4 weeks prior to the study
5. History of taking acupuncture

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The Questionnaire of Acupuncture Events | Every day during a 7 days trial

SECONDARY OUTCOMES:
Change from baseline on Mini-Mental State-Examination（MMSE）,The Behavioral Pathology in Alzheimer's Disease Rating Scale（BEHAVE-AD）and Activity of Daily Living Scale（ADL） | Baseline and 1week after the trial begen
Treatment Emergent Symptom Scale (TESS) | Baseline and 2 weeks after the trial begen

CONTACTS AND LOCATIONS:
Overall Officials: Yong Tang, M.D, Study Director — Chengdu University of TCM
Locations (1):
- Yong Tang, Chengdu, Sichuan, China